CLINICAL TRIAL: NCT05925439
Title: Comparison of the Incidence of Intravascular Injection Using the Tuohy and Quincke Needles During Ultrasound-guided S1 Transforaminal Epidural Injection: a Prospective Randomized Controlled Study
Brief Title: Comparison of Tuohy Needle and Quincke Needle During S1 Transforaminal Epidural Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Clinical assistant professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2023-0145
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: S1 Transforaminal Epidural Block

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuohy needle group (Experimental): Ultrasound-guided S1 transforaminal epidural block with Touhy needle
  Interventions: Device: Tuohy needle group
- Quincke needle group (Active Comparator): Ultrasound-guided S1 transforaminal epidural block with Quincke needle
  Interventions: Device: Quincke needle group

INTERVENTIONS:
Device: Tuohy needle group — Ultrasound-guided S1 transforaminal epidural block with Touhy needle
  Arms: Tuohy needle group
Device: Quincke needle group — Ultrasound-guided S1 transforaminal epidural block with Quincke needle
  Arms: Quincke needle group

SUMMARY:
Recently, Park et al. introduced a new technique for performing S1 TFESI using ultrasound. S1 TFESI using ultrasound can be considered to overcome the disadvantages of exposure to radiation. We hypothesized that the frequency of intravascular injection differs depending on the type of needle during S1 TFESI under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient diagnosed with S1 radiculopathy because S1 root compression was confirmed on MRI and related symptoms 2. NRS of back and/or radiating pain score of 4 or more 3. Patients aged 19 years or older

Exclusion Criteria:

* 1. Cases in which lumbar count is expected to be difficult due to lumbarization, sacralization, or lumbosacral transition 2. When the S1 posterior foramen is not clearly identified on ultrasound 3. Malignancy 4. Systemic infections 5. Bleeding tendency 6. Contrast allergy 7. Pregnant Women 8. If you cannot read or agree to the consent form 9. If you are unable to sign the consent form yourself

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-06-22 (Estimated); Study Completion 2025-06-22 (Estimated)

PRIMARY OUTCOMES:
incidence of intravascular injection | 1 minute after finishing the procedure
  incidence of intravascular injection during S1 transforaminal epidural block

SECONDARY OUTCOMES:
time required to complete S1 transforaminal epidural block | Baseline, 1 second after the completion of the procedure
  time required to complete S1 transforaminal epidural block

CONTACTS AND LOCATIONS:
Overall Officials: Do-Hyeong Kim, Principal Investigator — Yonsei University
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea